CLINICAL TRIAL: NCT02230124
Title: Magnetic Resonance Elastography in Hydrocephalus
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: National Institute for Biomedical Imaging and Bioengineering (NIBIB) (NIH)
Responsible Party: Principal Investigator, Keith D. Paulsen, Professor, Dartmouth-Hitchcock Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: DMS 20618 FED07029; 3R01EB004632-02 (NIH)
Record Dates: First submitted 2014-08-28; First posted 2014-09-03 (Estimated); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Hydrocephalus
Keywords: Hydrocephalus
MeSH Terms: conditions — Hydrocephalus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MRE (Experimental)
  Interventions: Device: MRE

INTERVENTIONS:
Device: MRE

SUMMARY:
The purpose of this project is to assess the utility of a new magnetic resonance technique called magnetic resonance elastography (MRE) in the non-invasive diagnosis of normal pressure hydrocephalus. The investigators hypothesize that MRE produces a unique imaging signature for hydrocephalus that distinguishes the disease from the normal (non-hydrocephalic) but atrophied brain, a distinction not possible with conventional MR imaging studies that are presently available.

ELIGIBILITY:
Inclusion Criteria:

* Age >21;
* One or more of the following complaints: memory loss/dementia, urinary incontinence, or progressive gait disturbance
* Ventriculomegaly defined as temporal horn width >2 mm or a FH:ID ratio>30% on computed tomography or MRI, where FH is the maximal distance between the frontal horns and ID is the internal diameter from inner table to inner table of the skull at this level (Greenberg)
* A diagnosis of any adult onset hydrocephalus (NPH, post-traumatic, post-hemorrhagic, obstructive, or idiopathic) will be considered for enrollment in this study

Exclusion Criteria:

* Implanted neuro-stimulator or cardiac pacemaker
* Known coagulopathy; major organ dysfunction
* End-stage congestive heart failure
* Oxygen-dependent pulmonary disease, hepatic cirrhosis, or dialysis- dependent renal failure; or other condition which, according to the assessment of the treating surgeon or anesthesia team
* Precludes consideration of elective surgery
* Patients who may be pregnant will be excluded from this study as well

Ages: 45 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2007-03-01 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Mean shear modulus | 15 Years
  The primary outcome measure will be mean shear modulus determined from pre-operative (and pre-drain placement) MRE in patients who demonstrate clinical improvement with trial CSF drainage versus patients who do not demonstrate improvement.

SECONDARY OUTCOMES:
Pre-operative (and pre-drain placement) shear modulus in the experimental group will be compared with various assessments of clinical improvement after VP shunting. | 15 Years
  Secondary outcomes will compare pre- and post-drain MRE shear moduli with ventricular size and intracranial pressure.

CONTACTS AND LOCATIONS:
Overall Officials: Keith D Paulsen, PhD, Principal Investigator — Dartmouth College
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States